CLINICAL TRIAL: NCT01919112
Title: Non-invasive Brain Stimulation for Swallowing Recovery After a Dysphagic Stroke
Brief Title: Fostering Eating After Stroke With Transcranial Direct Current Stimulation
Acronym: FEASt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Sandeep Kumar, Associate Professor of Neurology, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013P000067; 1R01DC012584-01A1 (NIH)
Record Dates: First submitted 2013-08-06; First posted 2013-08-08 (Estimated); Results first posted 2020-07-07 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Dysphagia; Stroke
Keywords: Brain stimulation
MeSH Terms: conditions — Deglutition Disorders; Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: The trial will randomize subjects to anodal transcranial direct current stimulation (tDCS) versus sham stimulation, both of them carried out in combination with standardized swallowing exercises
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigators and subjects will be masked to the trail arm assignments at randomization. The investigator reviewing outcome data will also be masked to the trial assignments.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High dose anodal tDCS (Experimental): High dose tDCS (2 milliamps twice daily) for 5 days will be administered concomitantly with swallowing exercises
  Interventions: Device: tDCS
- Low dose anodal tDCS (Active Comparator): This arm will use a low dose of current administered via tDCS (2 milliamps once daily) for 5 days will be administered concomitantly with swallowing exercises
  Interventions: Device: tDCS
- Sham Stimulation (Sham Comparator): Twice daily swallowing exercises only
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — Anodal tDCS will be administered with swallowing exercises

SUMMARY:
Swallowing difficulties are common after a stroke and can lead to serious complications like pneumonia and malnutrition. Unfortunately, there are no effective treatment for improving swallowing in stroke patients.

Previous investigations have shown that recovery of swallowing functions occurs from reorganization ("rewiring") of the non-involved cerebral hemisphere. In this study, the investigators propose to investigate a new intervention, which combines, swallowing exercises with brain stimulation targeted to the non-involved cerebral hemisphere, using low intensity current in acute stroke patients. The investigators plan to assess the safety of this technique in this patient population and also assess its effect on improving swallowing functions and swallowing physiology. During this time trial participants will undergo standardized swallowing and neurological assessments as well as brain MRI scans.

DETAILED DESCRIPTION:
Swallowing impairments are a common and a serious complication of stroke but lack effective therapies. The study investigators herein propose to conduct a prospective clinical study using a non-invasive brain stimulation technique, anodal transcranial direct current stimulation (tDCS), in combination with swallowing exercises for improving dysphagia due to an acute-subacute hemispheric infarction, and obtain data on safety and effect of 2 different doses of tDCS, on swallowing physiology and behavior. Dysphagia from hemispheric strokes occurs due to disruption of the cortical projections to the brainstem swallowing centers while recovery of swallowing functions have been shown to be mediated via the reorganization of the swallowing cortex in the unaffected hemisphere. A recent pilot study conducted by the investigators demonstrated the safety and feasibility of applying 5 consecutive daily sessions of anodal tDCS for 30 minutes to the swallowing cortex on the unaffected hemisphere in the acute-subacute stroke phases and showed a promise in improving dysphagia, when combined with swallowing exercises. The proposed research will be used to further confirm safety of this technique in early stroke phases and explore alternative, more effective doses for promoting swallowing recovery prior to its examination in any confirmatory trials. The investigators will use the study cohort to examine important subject specific parameters which influence response to the proposed intervention in dysphagic stroke patients. The overall aim of this study is to gather additional safety data on cumulative sessions of tDCS in acute-subacute phases of stroke, obtain information about effects of this intervention on important physiological and clinically relevant swallowing parameters, examine possible dose effects, and identify candidates who are more likely to benefit from this intervention. The experience gained from this project will guide planning of future confirmatory trials that use relevant clinical outcomes to assess potential benefits of this intervention and utilize important subject specific parameters to refine study inclusion criteria and aid in severity adjusted analysis.

ELIGIBILITY:
Inclusion Criteria:

* 21 years or older in age since safety of non-invasive cortical stimulation in children.
* Between 25 hours (day 2) to 144 (day 6) hours since stroke onset.
* Unilateral hemispheric infarction (cortical or subcortical infarction) documented by imaging.
* Moderate to severe dysphagia with a score of 4 or more on Penetration and Aspiration Scale (PAS)

Exclusion Criteria:

* Prior history of swallowing difficulties.
* Drowsiness or marked cognitive impairment that interferes with participation in swallowing maneuvers.
* Unable to undergo an MRI due to claustrophobia or presence of electrically, magnetically or mechanically activated implant (including cardiac pacemaker), intracerebral vascular clips or any other electrically sensitive support system, metal in any part of the body, including metallic injury to eye, or pregnancy).
* History of seizures or unexplained episodes of loss of consciousness.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Kumar, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Marchina S, Schlaug G, Kumar S. Study design for the fostering eating after stroke with transcranial direct current stimulation trial: a randomized controlled intervention for improving Dysphagia after acute ischemic stroke. J Stroke Cerebrovasc Dis. 2015 Mar;24(3):511-20. doi: 10.1016/j.jstrokecerebrovasdis.2014.09.027. Epub 2014 Dec 19. PMID 25534369

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects were recruited from the inpatient neurology/stroke service at Beth Israel Deaconess Medical Center, Boston, MA. The first subject was recruited on 2/10/2014.
Pre-assignment Details: A total of 328 subjects were screened for the trial, of which 214 did not fulfill all trial criteria and 72 refused consent. A total of 42 subjects were eventually enrolled: 14 subjects in High-Dose tDCS, 13 in Low-Dose tDCS and 15 in Sham arms.
Period: Primary Analysis-day 5 of Intervention
Arm/Group | High Dose Anodal tDCS | Low Dose Anodal tDCS | Sham Stimulation
Started | 14 | 13 | 15
Completed | 14 | 13 | 15
Not Completed | 0 | 0 | 0
Period: Secondary Analysis-day 30
Arm/Group | High Dose Anodal tDCS | Low Dose Anodal tDCS | Sham Stimulation
Started | 14 | 13 | 15
Completed | 12 | 12 | 14
Not Completed | 2 | 1 | 1
Not completed — Death | 1 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose Anodal tDCS | Low Dose Anodal tDCS | Sham Stimulation | Total
Number analyzed (Participants) | 14 | 13 | 15 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (12.6) | 72 (13.3) | 73 (14.1) | 71 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 8 | 6 | 17
  Male | 11 | 5 | 9 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 3
  Not Hispanic or Latino | 12 | 13 | 14 | 39
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 0 | 5
  White | 9 | 11 | 14 | 34
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 14 | 13 | 15 | 42
Penetration and Aspiration Scale Score [Mean (Standard Deviation); unit: units on a scale] — This is a validated 8 point ordinal scale (range 1-8; score 1 is normal and 8 is the worst possible) that quantifies penetration and aspiration events observed during a videofluroscopic swallowing study (VFSS). All PAS scores were assigned by an independent evaluator blinded to intervention allocation and were based on a standardized VFSS.
  units on a scale | 4 (1.2) | 4.1 (1.1) | 4 (1.5) | 4 (1.3)

OUTCOME MEASURES:

1. Primary Outcome: To Assess Changes in Penetration and Aspiration
Description: This will be assessed using the Penetration and Aspiration Scale (PAS) scores, a validated 8 point ordinal scale that quantifies penetration and aspiration events observed during Videofluoroscopic Swallowing Evaluation. PAS ranges from 1 (best score) representing no aspiration or penetration to 8 (worst score) representing severe aspiration. An average PAS score will be computed based on 9 swallows for this outcome.
Time Frame: Scores will be measured before tDCS and after 5 days after completion of stimulation
Population: Analysis of participant was based on an intention to treat principle.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Dose Anodal tDCS | Low Dose Anodal tDCS | Sham Stimulation
Number analyzed (Participants) | 14 | 13 | 15
score on a scale | -0.4 (1.2) | -0.8 (1.5) | -0.8 (1.6)

2. Primary Outcome: To Assess Safety of tDCS in Acute-subacute Stroke Phase: Number of Participants With Seizures in Each of the 3 Groups
Description: We will tabulate the number of participants who develop seizures in the High-dose anodal tDCS, Low-dose anodal tDCS and Sham stimulation groups.
Time Frame: During the 5 days of stimulation sessions
Population: Analyzed on an intention to treat as well as per protocol analysis
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Anodal tDCS | Low Dose Anodal tDCS | Sham Stimulation
Number analyzed (Participants) | 14 | 13 | 15
Participants | 0 | 0 | 0

3. Primary Outcome: To Assess Safety of tDCS in Acute-subacute Stroke Phase: Number of Deaths in Each of the 3 Groups Attributable to the Direct Effects of Stroke
Description: We will tabulate the number of deaths in High-dose tDCS, Low-dose tDCS and Sham stimulation groups, that are attributable to the direct effects of the qualifying stroke.
Time Frame: During the 5 days of stimulation sessions
Population: Analyzed on an intention to treat as well as per protocol analysis
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Anodal tDCS | Low Dose Anodal tDCS | Sham Stimulation
Number analyzed (Participants) | 14 | 13 | 15
Participants | 0 | 0 | 0

4. Primary Outcome: To Assess Safety of tDCS in Acute-subacute Stroke Phase: Number of Participants With Neurological Deterioration in Each of the 3 Groups
Description: We will tabulate the number of participants who develop neurological deterioration in the High-dose tDCS, Low-dose tDCS and Sham groups. Neurological deterioration will be defined as an increase in the total National Institute of Health Stroke Scale (NIHSS) Score by 4 or more points between each successive day. The NIHSS is a 15-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. NIHSS ranges from 0 (normal) to 42 (worst possible score). Higher scores mean worse neurological functions.
Time Frame: During the 5 days of stimulation sessions
Population: Analyzed on an intention to treat as well as per protocol analysis
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Anodal tDCS | Low Dose Anodal tDCS | Sham Stimulation
Number analyzed (Participants) | 14 | 13 | 15
Participants | 0 | 0 | 0

5. Primary Outcome: To Assess Safety of tDCS in Acute-subacute Stroke Phase: Number of Participants With Motor Deterioration in Each of the 3 Groups
Description: We will tabulate the number of participants with deterioration in their motor functions in the High-dose tDCS, Low-dose tDCS and Sham groups. Motor deterioration will be defined as an increase in the motor sub-item of the National Institute of Health Stroke Scale (NIHSS) score by 2 or more points between each successive day of stimulation. The motor sub-item of the NIHSS ranges from 0 (normal) to 16 (worst possible score), with higher scores indicating a worse motor exam.
Time Frame: During the 5 days of stimulation sessions
Population: Analyzed on an intention to treat as well as per protocol analysis
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Anodal tDCS | Low Dose Anodal tDCS | Sham Stimulation
Number analyzed (Participants) | 14 | 13 | 15
Participants | 0 | 0 | 0

6. Primary Outcome: To Assess Safety of tDCS in Acute-subacute Stroke Phase: Number of Participants With Swallowing Deterioration in Each of the 3 Groups
Description: We will tabulate the number of participants with swallowing deterioration in the High-dose tDCS, Low-dose tDCS and sham groups Swallowing deterioration will be defined as an increase in the score by 2 or more points in the Functional Oral Intake Scale (FOIS). FOIS provides a validated measure of diet level. FOIS is an ordinal scale ranging from 7 (normal diet) to 0 (no oral intake), with lower scores indicating a worse diet.
Time Frame: Any change between day 1 and day 3 of stimulation session
Population: Analyzed on an intention to treat as well as per protocol analysis
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Anodal tDCS | Low Dose Anodal tDCS | Sham Stimulation
Number analyzed (Participants) | 14 | 13 | 15
Participants | 0 | 0 | 0

7. Secondary Outcome: To Assess and Compare Changes in Dietary Intake in Each of the Three Groups
Description: The durability of any observed effects of the intervention on dietary status will be estimated by changes in Functional Oral Intake Scale (FOIS) score. FOIS is an ordinal scale ranging from 1 (worst) to 7 (normal oral diet) and provides a reliable measure of dietary intake. The change in FOIS scores across each group will be compared.
Time Frame: At study onset and after 1 month
Population: Analyzed on an intention to treat analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Dose Anodal tDCS | Low Dose Anodal tDCS | Sham Stimulation
Number analyzed (Participants) | 12 | 12 | 14
score on a scale | 2.9 (1.2) | 2.5 (1.7) | 2.1 (1.7)

8. Secondary Outcome: To Assess Changes in Physiological Measures of Pharyngeal Strength
Description: Examining effects of differing doses of anodal tDCS versus sham stimulation on Pharyngeal Constriction Ratio (PCR), derived from videofluoroscopic swallowing studies.PCR is a measure of the pharyngeal area visible in the lateral radiograph view at the point when a bolus is held in the oral cavity divided by the pharyngeal area at the point of maximum pharyngeal constriction during the swallow. A higher PCR indicates a weak swallow leading to increased food residue in the pharynx.
Time Frame: Variables will be measured at baseline (before starting tDCS) and after 5 days after completion of stimulation
Population: Analyzed on an intention to treat as well as per protocol analysis
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | High Dose Anodal tDCS | Low Dose Anodal tDCS | Sham Stimulation
Number analyzed (Participants) | 14 | 13 | 13
Ratio | -0.01 (0.09) | -0.1 (0.12) | -0.02 (0.06)

9. Secondary Outcome: To Assess Changes in Physiological Measures of Briskness of Swallow Onset
Description: Examining effects of differing doses of anodal tDCS versus sham stimulation on Pharyngeal Delay Time (PDT) , derived from videofluoroscopic swallowing studies. PDT is defined as the time in centiseconds that the bolus is present in the hypopharynx before the swallow is triggered. PDT is a temporal measure of the briskness of the swallow onset.
Time Frame: Variables will be measured at baseline (before starting tDCS) and after 5 days after completion of stimulation
Population: Analyzed on an intention to treat as well as per protocol analysis
Measure: Mean (Standard Deviation); unit: centiseconds
Arm/Group | High Dose Anodal tDCS | Low Dose Anodal tDCS | Sham Stimulation
Number analyzed (Participants) | 13 | 11 | 14
centiseconds | 5.2 (21.3) | -7.3 (43.4) | 0.83 (20.6)

10. Secondary Outcome: To Assess Changes in Physiological Measures of Laryngeal Excursion
Description: Examining effects of differing doses of anodal tDCS versus sham stimulation on measure of actual excursion of the larynx in centimeters from their resting point to maximal excursion, derived from videofluoroscopic swallowing studies.
Time Frame: Variables will be measured at baseline (before starting tDCS) and after 5 days after completion of stimulation
Population: Analyzed on an intention to treat as well as per protocol analysis
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | High Dose Anodal tDCS | Low Dose Anodal tDCS | Sham Stimulation
Number analyzed (Participants) | 12 | 9 | 12
centimeters | 0.07 (0.81) | 0.17 (1.4) | 0.14 (0.67)

11. Secondary Outcome: Change in PAS Scores as an Indicator of Dysphagia Recovery After Covariate Adjustment
Description: We will examine the effects of the intervention in a linear model by using it as a predictor for dysphagia recovery along with other variables of interest [age, baseline National Institute of Health Stroke Scale and Penetration and Aspiration Scale (PAS) scores], with a change in PAS scores from baseline to day 5 of the intervention, as being the outcome of interest.
Time Frame: At day 5 of study participation
Measure: Median (Standard Error); unit: score on a scale
Arm/Group | High Dose Anodal tDCS | Low Dose Anodal tDCS | Sham Stimulation
Number analyzed (Participants) | 14 | 13 | 15
score on a scale | -0.34 (0.35) | -0.81 (0.36) | -0.96 (0.33)
Statistical Analysis 1: Comparison: High Dose Anodal tDCS vs Low Dose Anodal tDCS vs Sham Stimulation; The aim for this analysis was to assess for effect modification of the trial intervention across the novel radiological variable corticobulbar tract-lesion load; Test type: Other — Regression models using interaction terms will used to assess for heterogeneity of intervention effects across the novel radiological variable corticobulbar tract (CBT)-lesion load, a combined measure of lesion size and location. For purposes of the analysis, the CBT-lesion load was dichotomized into 2 groups based on the median CBT-lesion load volume; p = 0.116, 2-way analysis of variance with interact — Interaction p-values will be considered statistically significant at the 0.15 level of significance given the relatively low power for tests of interaction to detect a true interaction; The tDCS intervention was the main variable of interest, PAS score the main outcome and CBT-lesion load was the interaction term used

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the entire duration of patient follow-up (30 days since trial enrollment).
Arm/Group | High Dose Anodal tDCS | Low Dose Anodal tDCS | Sham Stimulation
All-Cause Mortality (participants affected / at risk) | 1/14 | 1/13 | 1/15
Serious Adverse Events (participants affected / at risk) | 1/14 | 1/13 | 2/15
Other Adverse Events (participants affected / at risk) | 3/14 | 2/13 | 3/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Anodal tDCS (N=14) | Low Dose Anodal tDCS (N=13) | Sham Stimulation (N=15)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Anodal tDCS (N=14) | Low Dose Anodal tDCS (N=13) | Sham Stimulation (N=15)
Fever (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
hyperglycemia (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Metabolic disorder (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-08-14): https://cdn.clinicaltrials.gov/large-docs/12/NCT01919112/Prot_SAP_000.pdf